CLINICAL TRIAL: NCT05236101
Title: Validation of Child Drawing Hospital Scale (CD: H) and the Place of the Drawing in the Evaluation of Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halenur Altan, Assoc. Dr., Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-KAEK-195
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Dental Anxiety; Dental Pain; Validation; Child Drawing Hospital Scale
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD:H Scale (Experimental): Pictures drawn using the CD:H Scale were evaluated.
  Interventions: Behavioral: survey research

INTERVENTIONS:
Behavioral: survey research — Children with dental treatment were asked to draw pictures.

SUMMARY:
Objectives: Our study aimed to perform a Turkish validation study of the Child Drawing: Hospital (CD:H) Scale and evaluate the dental anxiety and pain experienced during the treatment by drawing.

Study Design: Pediatric patients between the ages of 4-13 who applied to the Pediatric Dentistry Department between 2018-2020 were included in the study. Following the translation of the CD:H Scale into Turkish and linguistic-cultural validation, the behaviors of pediatric patients during treatment were evaluated with the Frankl Behavior Rating Scale, the pain they experienced during treatment with the Wong- Baker Face Rating Scale, and their anxiety levels were evaluated with the pictures drawn by the patients at the end of the treatment. The data were analyzed with Statistical Package for the Social Sciences v23, and the significance level was taken as p <0.05.

Results: Within the scope of the scale's reliability-validity study, the Intra-Class Correlation Coefficient (ICC) was evaluated with test-retest consistency. For section A,B,C and total score reliability was found to be positive and strong level correlation. Dental anxiety of boys was higher than girls.

Conclusions: The Turkish version of the CD:H Scale is a reliable and valid scale that can be used to evaluate the dental anxiety of Turkish pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have toothache and who have undergone dental treatment (filling and root canal treatment)
* Patients with deep dentin caries who need local anesthesia
* Children between the ages of 4-13
* Patients who are willing to paint and understand commands
* Patients without any mental or physical disability
* Patients whose parents agreed to participate in the study and signed their consent

Exclusion Criteria:

* Children not aged 4-13
* Patients with mild to moderate caries who do not need local anesthesia
* Patients who are not willing to paint
* Patients with inadequate hand coordination
* Patients with motor dysfunction
* Children with any systemic illness
* Patients with mental or physical disabilities
* Patients with any syndrome
* Patients with color blindness
* Children whose native language is not Turkish
* Patients whose parents refused to participate in the study

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 235 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Turkish Validation of the Child Drawing Hospital Scale | 12 week
  Using the Child Drawing Hospital Scale, the pictures drawn by the patients were interpreted and scored by two researchers (minimum 15, max 205).

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozdemir Celik DS, Deniz E, Demir O, Altan H. Validation of child drawing hospital (CD: H) scale and the role of drawing in the evaluation of Dental anxiety. BMC Oral Health. 2025 Feb 21;25(1):274. doi: 10.1186/s12903-025-05605-2. PMID 39984891